CLINICAL TRIAL: NCT00156637
Title: A Study of Strategies to Improve Schizophrenia Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: MNT 02-210
Record Dates: First submitted 2005-09-07; First posted 2005-09-12 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2008-04

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: schizophrenia; quality of health care; quality indicators; intervention studies
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Other)
  Interventions: Behavioral: Team-Based Quality Improvement Intervention; Behavioral: Team Based Quality Improvement
- Arm 2 (Active Comparator): Dosing & Side Effect Monitoring
  Interventions: Behavioral: Opinion Leader Intervention

INTERVENTIONS:
Behavioral: Team-Based Quality Improvement Intervention — Intervention to improve recommended dosing and side effect monitoring of antipsychotic medications using a team-based quality improvement effort
  Arms: Arm 1
Behavioral: Opinion Leader Intervention — Intervention to improve recommended dosing and side effect monitoring of antpsychotic medications using an Opion leader quality improvement effort
  Arms: Arm 2
Behavioral: Team Based Quality Improvement — Intervention to increase appropriate use of clozapine through a team based quality intervention.
  Arms: Arm 1

SUMMARY:
The goal of this project is to translate research findings about key aspects of antipsychotic treatment into routine care through a multi-component intervention, focusing on improving two aspects of medication management that are directly linked to patient outcomes: 1) monitoring for potentially serious metabolic side effects of newer antipsychotic medication, and 2) increasing the appropriate use of clozapine for treatment-refractory patients.

DETAILED DESCRIPTION:
Background:

Antipsychotic medication is by far the most widely utilized treatment for schizophrenia in VA settings, and the VA has established guidelines for the appropriate use of these medications. The recent introduction of a new generation of antipsychotic medications has also offered great hope to persons with schizophrenia, but also may adversely affect health due to metabolic side effects. Improving all aspects of antipsychotic medication management is necessary to improve outcomes for persons with schizophrenia.

Objectives:

The goal of this project is to translate research findings about key aspects of antipsychotic treatment into routine care through a multi-component intervention. Mental Health QUERI's (MHQ) previous project for improving antipsychotic treatment demonstrated that a multi-component intervention improved use of guideline-recommended antipsychotic doses. This project will build on results and lessons learned from MHQ's previous translation project. The scope of translation will be expanded from an ongoing focus on reducing high antipsychotic doses to include two additional aspects of medication management that are directly linked to patient outcomes: 1) increasing monitoring for potentially serious side effects of newer antipsychotic medication, and 2) increasing the appropriate use of clozapine for treatment-refractory patients.

Methods:

The project is employing a multi-component intervention for improving antipsychotic prescribing while comparing the use of two different interpersonal marketing/influence strategies for translation. The primary objective is to compare the effectiveness of a team-based QI approach and a strategy using a clinical opinion leader augmented by an implementation coordinator to improve antipsychotic medication management. In addition, MHQ will determine the impact of a support and consultation program to promote clozapine prescribing. A total of ten VA Medical Centers from 4 different VA health care networks (VISNs) have been selected to participate on the basis of number of patients with schizophrenia, baseline performance on quality indicators, and organizational characteristics. Six of these sites will focus on side effect monitoring and antipsychotic dosing (two team-based QI, two clinical opinion leader, and two control), while two will receive the clozapine consultation program, with two matched control sites. Selected clinicians and staff (opinion leaders) will be identified and trained, and will implement the multi-component intervention consisting of educational materials and programs, information system tools, and performance monitoring and feedback. The intervention will take place for 6 months, and will be assessed with regard to improvement in side effect monitoring, high dose antipsychotic prescribing, and clozapine use. In addition, MHQ will assess impact of the intervention on patient outcomes at five of the sites.

Status:

In partnership with clinical stakeholders, the project team is implementing, adapting and evaluating an assortment of clinical tools and training materials designed to improve antipsychotic medication management. All, sites, except 1, have completed the intervention. All subject recruitment had been completed. The project team is also working with participating VAMC IT staff and Clinical Coordinators to fully automate the project's VISTA data extraction reoutines and performance monitoring reporting system for local implmentation and maintainence

ELIGIBILITY:
Inclusion Criteria:

SITE: 300 or more patients with schizophrenia diagnosis Below national VA average on high antipsychotic dosing (dosing sites) or use of clozapine (clozapine sites)?Site leader buy-in

PATIENT: Clinical diagnosis of schizophrenia or schizoaffective disorder

18-65 years of age Had at least 1 inpatient stays or outpatient visits to facility in past year [Dosing Sites] Filled antipsychotic prescription at dose that exceeds guideline recommendations in past 3 months [Clozapine Sites] Scores positive on computer routine to identify potential candidates for a trial of clozapine

Exclusion Criteria:

SITE:No affiliation with an Institutional Review Board or Research and Development office for protocol review/approval PATIENT: No access to telephone Enrolled in a conflicting study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2005-06; Primary Completion 2007-01 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Antipsychotic dose above guideline-recommended range Side effect monitoring 30 days before/after new antipsychotic Clozapine prescribing for treatment-refractory schizophrenia | 6 months

SECONDARY OUTCOMES:
Patient functional status ?Improvement in schizophrenia symptoms Service Use

CONTACTS AND LOCATIONS:
Overall Officials: Richard R. Owen, MD, Principal Investigator — Central Arkansas Veterans Healthcare System Eugene J. Towbin Healthcare Center, Little Rock, AR
Locations (4):
- United States (4):
  - Veterans Health Care System of the Ozarks, Fayetteville, AR, Fayetteville, Arkansas
  - Central Arkansas Veterans Healthcare System Eugene J. Towbin Healthcare Center, Little Rock, AR, No. Little Rock, Arkansas
  - Dayton VA Medical Center, Dayton, OH, Dayton, Ohio
  - Michael E. DeBakey VA Medical Center, Houston, TX, Houston, Texas

REFERENCES:
- [Result] Rosen CS, Tiet QQ, Harris AH, Julian TF, McKay JR, Moore WM, Owen RR, Rogers S, Rosito O, Smith DE, Smith MW, Schnurr PP. Telephone monitoring and support after discharge from residential PTSD treatment: a randomized controlled trial. Psychiatr Serv. 2013 Jan;64(1):13-20. doi: 10.1176/appi.ps.201200142. PMID 23117443
- [Result] Young AS, Niv N, Chinman M, Dixon L, Eisen SV, Fischer EP, Smith J, Valenstein M, Marder SR, Owen RR. Routine outcomes monitoring to support improving care for schizophrenia: report from the VA Mental Health QUERI. Community Ment Health J. 2011 Apr;47(2):123-35. doi: 10.1007/s10597-010-9328-y. Epub 2010 Jul 25. PMID 20658320